ID: RE16-00001 Clinical Follow-up of Anti-Carbamylated Antibody NCT02958319 Status in Rheumatoid Arthritis

Date of document: November 25th, 2021

## **Study Statistical Methods**

We will use descriptive statistics for categorical and numerical variables. Categorical variables will be expressed in frequency and percentage; comparisons will be done by chi square test. Numerical variables, after normality test will be described as mean and median with SD and IQR, respectively.

For the primary end point we will compare by chi square test the percentage of DAS28-VSG remission by group.

For the secondary endpoints we will compare by t test or U Mann Whitney the mean o median of the cumulative dose of prednisone and number of DMARDs used.